CLINICAL TRIAL: NCT00597220
Title: Randomized, Prospective, Placebo-controlled, Multi-center Study to Test the Efficacy of n-3 PUFA for the Maintenance of Normal Sinus Rhythm in Patients With Persistent Atrial Fibrillation
Brief Title: Randomized Trial to Assess Efficacy of PUFA for the Maintenance of Sinus Rhythm in Persistent Atrial Fibrillation
Acronym: FORWARD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacion GESICA (Other)
Responsible Party: Alejandro Macchia, Fundacion GESICA
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FORWARD
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Omega 3
  Interventions: Dietary Supplement: Omega 3 (n-3 PUFA)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Omega 3 (n-3 PUFA) — 1 gram of n-3 PUFA containing DHA and EPA
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
To demonstrate that in patients with persistent atrial fibrillation who had recovered normal sinus rhythm and treated with the best recommended therapies, the addition of 1 gram / daily of n-3 PUFA is superior to the corresponding placebo for the maintenance of normal sinus rhythm at one year of follow up.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) impose a substantial and growing economic burden on health care expenditures. In patients with persistent AF, there are fundamentally two ways to manage the arrhythmia: to restore and maintain sinus rhythm (rhythm control) or to allow AF to continue and ensure that the ventricular rate is controlled (rate control). As it has been stated, it goes without saying that if we could prevent atrial fibrillation (AF) or restore and maintain sinus rhythm in patients suffering from persistent AF, without any penalties due to the unwanted effects of drugs or incomplete suppression of AF and its thromboembolic complications, every physician would do so. Current strategies however, are limited to achieve such desirable goal. In the last years a growing amount of evidence and attention regarding the cardio-protective role of Omega 3 fatty acids (n-3 PUFA) became progressively clear and appealing.

Epidemiological studies and randomized controlled trials confirms the role of n-3 PUFA in reducing all cause mortality and cardiovascular events mostly in patients at high cardiovascular risk. These effects seems to be mediated mostly by an anti-arrhythmogenic effect.

Basic science confirms and extended clinical observations regarding the antiarrhythmogenic effect of these compounds. Recently both basic research and clinical science suggested a role of n-3 PUFA for the prevention and treatment of supraventricular arrhythmias, particularly AF.

The purpose of the study is to show that the addition of n-3 PUFA on the top of the best recommended therapies can improve the maintenance of normal sinus rhythm in patients with persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Persistent atrial fibrillation

Exclusion Criteria:

* Contraindications or known hypersensitivity to n-3 PUFA
* Current treatment with n-3 PUFA for any reason
* Heart failure NYHA class IV
* Coronary artery bypass surgery or valve replacement within the past 3 months
* Planned cardiac procedures
* Known sick-sinus syndrome
* Diagnosis of Wolff-Parkinson-White
* Clinical significant valvular etiologies
* Presence of arrhythmia associated with an acute reversible condition
* Advanced chronic lung disease
* Contraindications for anticoagulation therapy
* Pregnancy or lactation
* Any non cardiac illness associated with a life expectancy of < 2 years
* Treatment with any investigational agent within 3 month before randomization
* Any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety or be associated with poor adherence to the protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-07 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Survival free of atrial fibrillation | 12 months

SECONDARY OUTCOMES:
Number of patients in sinus rhythm at the time of each study visit | 12 months
Number of hospitalizations for CV reasons | 12 months
Number of all-cause hospitalizations | 12 months
Incidence of TE events | 12 months
Number of patients who die or with non-fatal thromboembolic events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hernan C Doval, MD, Study Chair — Fundacion GESICA; Gianni Tognoni, MD, Study Chair — Mario Negri Institute; Hugo Grancelli, MD, Study Director — Fundacion GESICA; Sergio Varini, MD, Study Director — Fundacion GESICA; Daniel Nul, MD, Study Director — Fundacion GESICA; Alejandro Macchia, MD, Study Director — Fundacion GESICA
Locations (13):
- Argentina (13):
  - Hospital Alemán, Caba, Buenos Aires
  - Clinica Constituyentes, Caba, Buenos Aires
  - Complejo Medico Policial Churruca Visca, Caba, Buenos Aires
  - Fundacion Favaloro, Caba, Buenos Aires
  - Hospital Evita Pueblo FEDITEC, Lanús, Buenos Aires
  - Clinica y Maternidad Colon, Mar del Plata, Buenos Aires
  - Hospital Privado de la Comunidad, Mar del Plata, Buenos Aires
  - Hospital José de San Martín, Corrientes, Corrientes Province
  - Clinica Romagosa, Córdoba, Córdoba Province
  - Sanatorio Integral IOT, Misiones, Misiones Province
  - Centro Cardiovascular Salta, Salta, Salta Province
  - Sanatorio Parque, Rosario, Santa Fe Province
  - CEMIC (Centro de Educación Médica e Investigaciones Clinicas Norberto Quirno), Buenos Aires

REFERENCES:
- [Derived] Macchia A, Grancelli H, Varini S, Nul D, Laffaye N, Mariani J, Ferrante D, Badra R, Figal J, Ramos S, Tognoni G, Doval HC; GESICA Investigators. Omega-3 fatty acids for the prevention of recurrent symptomatic atrial fibrillation: results of the FORWARD (Randomized Trial to Assess Efficacy of PUFA for the Maintenance of Sinus Rhythm in Persistent Atrial Fibrillation) trial. J Am Coll Cardiol. 2013 Jan 29;61(4):463-468. doi: 10.1016/j.jacc.2012.11.021. Epub 2012 Dec 19. PMID 23265344
- [Derived] Macchia A, Varini S, Grancelli H, Nul D, Laffaye N, Ferrante D, Tognoni G, Doval HC; FORomegaARD investigators. The rationale and design of the FORomegaARD Trial: A randomized, double-blind, placebo-controlled, independent study to test the efficacy of n-3 PUFA for the maintenance of normal sinus rhythm in patients with previous atrial fibrillation. Am Heart J. 2009 Mar;157(3):423-7. doi: 10.1016/j.ahj.2008.10.027. Epub 2009 Jan 8. PMID 19249410